CLINICAL TRIAL: NCT03547076
Title: The Use of Handheld Ultrasound Utilizing Support by Experts or Automatic Analyses for Improved Diagnostics at Remote Locations
Brief Title: Handheld Ultrasound at Remote Locations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Norwegian University of Science and Technology (Other); Levanger and Verdal Muncipality (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: LE-2018_GP1
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure
Keywords: Pocket sized imaging device; Handheld ultrasound device; General practitioner; Nurse; Focused cardiac ultrasound; FoCUS; Telemedicine; Support
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The focused Pocket ultrasound examination and evaluation will be performed by a general practitioner. A similar focused ultrasound examination will be performed by a nurse without evaluation by the nurse. The complete echocardiographic examination by a cardiologist, using a state of the art ultrasound machine is considered the gold standard method.
Masking Description: All study personnel will be masked for findings by other study personnel. Patients will first be examined by nurses or GP in a random order, then subsequently, reference examination will be performed by cardiologist experienced in heart failure diagnostics and echocardiography.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Focused ultrasound diagnostics (Experimental): Intervention: Focused ultrasound Diagnostics
  All participants will first be examined twice with handheld ultrasound, With separate examinations performed by general practioners and nurses (random order). Both will utilize automatic analyses of left ventricular function and telemedicine support for best possible diagnosis of heart failure. Subsequently, reference imaging and diagnostics will be performed by experts (cardiologists). Handheld ultrasound examinations will be compared to Reference.
  Interventions: Diagnostic Test: Focused ultrasound diagnostics

INTERVENTIONS:
Diagnostic Test: Focused ultrasound diagnostics — Patients first be examined by nurses using a pocket-sized imaging device. Secondly, by a General Practitioner using the pocket-sized imaging device. Thirdly, reference echocardiography will be performed by cardiologist using a high-end echocardiographic scanner. Only tools (ultrasound equipment and dedicated software) approved for clinical practice will be used.
  The focused ultrasound examination includes three standard apical views (4-chamber, 2-chamber and long axis) with and without color Doppler, in addition to recordings from both pleural cavities and the inferior vena cava. The reference imaging includes the same recordings, but in addition all other chambers and valves are assessed (grey scale, color Doppler, pulsed wave and continuous wave Doppler and tissue Doppler).

SUMMARY:
Heart failure causes a large patient and financial burden on the health care system. Pocket ultrasound imaging devices are utilized to improve time to correct diagnosis. Telemedicine is used in a variety of medical professions today. A combination of focused handheld ultrasound imaging performed by general practitioners and dedicated nurses in a heart failure population, utilizing telemedicine for support, has not yet been studied. The aim of the study is to evaluate the feasibility, reliability and clinical influence of implementing handheld focused cardiac ultrasound by general practitioners and nurses for diagnostics and health-related expenditure in outpatients referred with suspected heart failure.

DETAILED DESCRIPTION:
Handheld focused cardiac ultrasound in diagnosis of suspected heart failure

Diagnostic ultrasound is more frequently used by clinicians in different scenarios. Echocardiography (cardiac ultrasound) is the most frequently method used when diagnosing heart failure (HF), cardiomyopathies, valvular pathology and cardiac tamponade, as well as other diseases affecting the heart, great vessels and pleural cavity. Ideally, the diagnostic workflow should conclude with a correct diagnosis as soon as possible, as this is important for preserving health and quality of life for the patients, as well as for total health care expenditure and the diagnostic workflow logistics.

For the last 6-7 years smaller and cheaper ultrasound scanners have become available. These pocket-sized (or handheld) imaging devices (PSIDs) have allowed for more inexperienced users, at locations outside the dedicated ultrasound laboratories, to perform ultrasound diagnostics. PSIDs fits in the "white coat" pocket and may be brought to the patient, and thus, allowing diagnostic imaging examinations to be performed at the patients' point-of-care. PSIDs from different vendors are available on the market. Large efforts are made in developing dedicated software helping the inexperienced users to maximize the diagnostic gain of including PSIDs in the diagnostic workflow. Experts have launched the PSIDs as the next generation stethoscope.

The cardiac research groups at Levanger Hospital and NTNU (Norway) have recently evaluated the PSID Vscan® from GE Ultrasound in several studies where the PSID has been tested on cardiac patients by different users. The PSID allow for improved diagnostics by both experts, residents, general practitioners (GPs), as well as medical students and dedicated nurses.

In the inpatients setting the population is selected and the prevalence of disease is high. Research has shown that by using the PSIDs the diagnosis was corrected in up to 1 of 5 medical inpatients. With less experienced users the diagnostic impact may be reduced. Studies from outpatient hospital settings have shown that the PSIDs may allow for diagnostic gain both in cardiac and non-cardiac care. Studies evaluating the influence of using PSIDs by GPs or other health care personnel outside the hospitals are scarce. Thus, there is a need for studies evaluating the use of PSIDs or other imaging modalities performed by the GPs in the outpatient setting.

Education

For all inexperienced users, that are non-experts, dedicated training and education is mandatory to optimize gain and minimize misdiagnosis and subsequent imaging procedures. The gain of including PSIDs in the diagnostic workflow largely depends on the population examined. In the latest recommendation from the European Association of Cardiovascular Imaging (EACVI) no specific numbers are given for the training program, neither regarding time nor number of examinations. However, it is stated that "since the competency in FoCUS (Focused Cardiac UltraSound) should be the minimal net result of the training process, the number of required hours/studies might be adjusted for each trainee according to the results of the competency evaluation incorporated into the ongoing training process". The training program should aim to educate the user in the specific use of the PSIDs relevant for the planned scenarios to "ensure that the operators are aware of their own capacity and limitations, given the specific equipment and different situations".

Telemedicine The health care system of today has implemented a variety of technical tools that are based on advanced technological innovations. Such advances usually require highly technical and medical skills of the users, for optimization of the use and outcome of the advances. The advances in information technology, communication bandwidth capacities of both wired and non-wired networks have made the basis for performing the diagnostics at one place and interpret the diagnostic tests at another location. According to the World Health Organization, telemedicine is defined as "the delivery of health care services, where distance is a critical factor, by all health care professionals using information and communication technologies for the exchange of valid information for diagnosis, treatment and prevention of disease and injuries, research and evaluation, and for the continuing education of health care providers, all in the interests of advancing the health of individuals and their communities".

Telemedicine has among others been implemented in radiology, where teleradiology is a common and accepted form in the diagnostic process. The methodology was first implemented in clinical scenarios where the need for a physical meeting between the patient and the physician was lower than the need for the specific tests. Traditionally, ultrasound examinations have been performed by highly specialized personnel and interpreted by the specialist more or less real time and at the same location.

User support Technological advances with the invention of easy-to-use, cheap and attainable ultrasound devices has allowed for a broader spectrum of users to implement ultrasound diagnostics. From the health care providers' point of view, this may allow for moving diagnostics to the patients' point-of-care, in contrast to moving the patients to the diagnostic laboratories. To implement ultrasound diagnostics outside the dedicated diagnostics laboratories, education and support of the users is mandatory. Even though inexperienced users easily can be trained to perform ultrasound images with indices, the interpretation of the images of anatomical structures and cardiac function indices requires experience.

The more inexperienced users can be supported in different ways. Beyond the obligatory theoretical support by literature and possibility to discuss findings with experts, there is need for qualitative feedback on the ultrasound recordings. Telemedicine may offer secure transmission of the ultrasound recordings for interpretation by experts and allowing for discussion as well. The outpatient ultrasound recordings may also be included in hospital referrals. In addition, our research group has been involved in development of an algorithm which can automatically interpret ultrasound recordings of the function of the left ventricle. Such software can give quick feedback which may be helpful for training and education of the user, as well its possibility to improve the diagnostic ability of the ultrasound examination performed by the inexperienced user.

Heart failure Heart failure (HF) affects 15 million Europeans; incidence in Norway is 11.000 per year. The prevalence is increasing due to improvements in diagnostics and therapy, not to mention the increased age of the population. Health care expenditure related to management of heart failure is significant, both with respect to the financial costs and patient burden. Thus, early and correct diagnosis is important to improve patient care and reduce the financial burden on the health care system. Heart failure patients often have comorbidities, and hospitalization is common if not optimally monitored and treated. Today approximately 50% of heart failure patients are readmitted within 6 months after hospitalization for decompensated heart failure.

Hyper- and hypovolemia can both lead to decompensated HF and secondary organ failure caused by inadequate perfusion. However, pleural effusion is easy assessable by ultrasound and in a recent study we found that pleural effusion was present in 42% of the patients. Non-cardiologists may have a growing role in diagnostics and follow-up of outpatient HF patients, and adding ultrasound diagnostics to the consultations may improve care.

Telemedicine in follow-up of patients with chronic heart failure The most advanced way of monitoring chronic HF patients by telemedicine is the use of implantable devices for haemodynamic monitoring, where invasive pressures were automatically uploaded from implanted devices through a patient home monitoring system and used to guide treatment. The Remote monitoring has become appealing, and is a potentially cost-effective method of home management and prevention of readmission.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the outpatient clinic at Levanger Hospital for echocardiography due to suspicion of heart failure, which have consented to participate in the study.
* N-terminal pro brain natriuretic peptide (NT-proBNP) ≥125 ng/L or brain natriuretic peptide ≥35 ng/L

Exclusion Criteria:

* The patient is not able to consent.
* The patient has know heart failure
* Known result of any of the following cardiac imaging tests (echocardiography, cardiac magnet resonance imaging (MRI), cardiac (not coronary) computed tomography (CT).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical influence of diagnostic ultrasound examinations supported by telemedicine | Clinical influence will be tested on day 0 (time of study inclusion)
  Clinical influence will be evaluated by the proportion of patients correct evaluated to have or not to have heart failure by the use of handheld ultrasound

SECONDARY OUTCOMES:
Feasibility of handheld cardiac ultrasound performed by general practitioners | Feasibility will be tested on day 0 (time of study inclusion)
  ReliabiFeasibility, as the proportion of recordings, of cardiac ultrasound images allowing for assessment of left ventricular function by the operator.

OTHER OUTCOMES:
Feasibility of handheld cardiac ultrasound performed by general practitioners supported by automatic interpretation of left ventricular function. | Feasibility will be tested on day 0 (time of study inclusion)
  Feasibility, as the proportion of recordings, of cardiac ultrasound images allowing for assessment of left ventricular function by the algorithms included in the handheld ultrasound device. Specified will we evaluate the proportion of exams that is successfully recorded by the general practitioners and successfully automatically interpreted
Feasibility of handheld cardiac ultrasound performed by general practitioners with expert support by telemedicine | Feasibility will be tested on day 0 (time of study inclusion)
  Feasibility, as the proportion of recordings, of cardiac ultrasound images allowing for assessment of left ventricular function by the algorithms included in the handheld ultrasound device. Specified will we evaluate the proportion of exams that is successfully recorded by the general practitioners and successfully interpreted by experts utilizing a near real-time telemedicine approach.
Reliability of handheld cardiac ultrasound performed by general practitioners | Reliability will be tested on day 0 (time of study inclusion)
  Reliability, as the proportion of recordings, of cardiac ultrasound images allowing for assessment of left ventricular function by the operator.
Reliability of handheld cardiac ultrasound performed by general practitioners supported by automatic interpretation of left ventricular function. | Reliability will be tested on day 0 (time of study inclusion)
  Reliability (accuracy) will be tested with C-statistics of ultrasound performed by nurses at an outpatient heart failure clinic, with interpretation of left ventricular function by the algorithms included in the handheld ultrasound device compared to Reference imaging by specialists in cardiology
Reliability of handheld cardiac ultrasound performed by general practitioners with expert support by telemedicine | Reliability will be tested on day 0 (time of study inclusion)
  Reliability (accuracy) will be tested with C-statistics of ultrasound performed by nurses at an outpatient heart failure clinic, with interpretation by telemedicine support of cardiologist compared to Reference imaging by specialists in cardiology
Feasibility of handheld cardiac ultrasound performed by nurses supported by automatic interpretation of left ventricular function. | Feasibility will be tested on day 0 (time of study inclusion)
  Feasibility, as the proportion of recordings, of cardiac ultrasound images allowing for assessment of left ventricular function by the algorithms included in the handheld ultrasound device. Specified will we evaluate the proportion of exams that is successfully recorded by the nurses and successfully automatically interpreted
Feasibility of handheld cardiac ultrasound performed by nurses with expert support by telemedicine | Feasibility will be tested on day 0 (time of study inclusion)
  Feasibility, as the proportion of recordings, of cardiac ultrasound images allowing for assessment of left ventricular function by the algorithms included in the handheld ultrasound device. Specified will we evaluate the proportion of exams that is successfully recorded by the nurses and successfully interpreted by experts utilizing a near real-time telemedicine approach.
Reliability of handheld cardiac ultrasound performed by nurses supported by automatic interpretation of left ventricular function. | Reliability will be tested on day 0 (time of study inclusion)
  Reliability (accuracy) will be tested with C-statistics of ultrasound performed by nurses at an outpatient heart failure clinic, with interpretation of left ventricular function by the algorithms included in the handheld ultrasound device compared to Reference imaging by specialists in cardiology
Reliability of handheld cardiac ultrasound performed by nurses with expert support by telemedicine | Reliability will be tested on day 0 (time of study inclusion)
  Reliability (accuracy) will be tested with C-statistics of ultrasound performed by nurses at an outpatient heart failure clinic, with interpretation by telemedicine support of cardiologist compared to Reference imaging by specialists in cardiology
Time use of handheld cardiac ultrasound performed by inexperienced users with expert support by telemedicine | Time consumption will be tested on day 0 (time of study inclusion)
  Time used for the sum of recording of cardiac ultrasound examination, telemedicine transfer of recordings and telemedicine interpretation by experts.
Quality of cardiac ultrasound performed by general practitioners | Quality will be tested on day 0 (time of study inclusion)
  Evaluation of the quality of recordings of cardiac ultrasound obtained by the general practitioners as a semiquantitative score reflecting the whole examination compared to the reference images by the cardiologist.
Quality of cardiac ultrasound performed by nurses | Quality will be tested on day 0 (time of study inclusion)
  Evaluation of the quality of recordings of cardiac ultrasound obtained by the nurses as a semiquantitative score reflecting the whole examination compared to the reference images by the cardiologist.
Evaluation of different methods for cardiac ultrasound user support | Usability of methods of support will be tested on day 0 (time of study inclusion)
  User evaluation of the usability assessed by the system usability scale.
Health care related cost of diagnostic handheld ultrasound algorithms in patients with suspected heart failure examinations supported by telemedicine | Health care related cost will be tested on day 0 (time of study inclusion)
  Health care related cost will be evaluated by the costs related to the diagnostic algorithms in patients with suspected heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Havard Dalen, MD, PhD, Study Chair — Norwegian University of Science and Tehnology
Locations (1):
- Department of Medicine, Levanger Hospital, Nord-Trøndelag Health Trust, Levanger, Norway

IPD SHARING:
Plan to Share IPD: Undecided
IPD share will follow regulations from the institutions.

REFERENCES:
- [Derived] Hjorth-Hansen AK, Magelssen MI, Andersen GN, Graven T, Kleinau JO, Landstad B, Lovstakken L, Skjetne K, Mjolstad OC, Dalen H. Real-time automatic quantification of left ventricular function by hand-held ultrasound devices in patients with suspected heart failure: a feasibility study of a diagnostic test with data from general practitioners, nurses and cardiologists. BMJ Open. 2022 Oct 13;12(10):e063793. doi: 10.1136/bmjopen-2022-063793. PMID 36229153